CLINICAL TRIAL: NCT01783730
Title: Special Investigation in Japanese Rheumatoid Arthritis Patients Who Have no Previous Use of DMARDs and Biological Agents
Brief Title: Assessment of the Safety of Adalimumab in Rheumatoid Arthritis Patients Showing Rapid Progression of Structural Damage of the Joints, Who Have no Prior History of Treatment With Disease-modifying Anti-rheumatic Drugs or Biological Agents
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-983
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with high rheumatoid arthritis disease activity: Participants who received adalimumab treatment

SUMMARY:
This study was conducted to examine the safety profile and the effectiveness in daily clinical practice of adalimumab in rheumatoid arthritis participants showing rapid progression of structural damage of the joints, who had no prior history of treatment with disease-modifying anti-rheumatic drugs or biological agents.

DETAILED DESCRIPTION:
This was a multicenter, prospective, observational study of adalimumab. Each participant enrolled when initiating adalimumab treatment and was to be followed up for 24 weeks or until discontinuation of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. High disease activity, with poor prognostic factors (e.g., rheumatoid factor [RF]-positive, anti-cyclic citrullinated peptide [CCP] antibody-positive, or bone erosion)
2. Combination of adalimumab and methotrexate will be started
3. No prior history of treatment with disease-modifying anti-rheumatic drugs
4. No prior history of treatment with biological agents
5. Adalimumab dosed according to the registered product label
6. Signed informed consent

Exclusion Criteria:

There were no specific exclusion criteria.

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rheumatoid Arthritis participants showing rapid progression of structural damage of the joints, who have no prior history of treatment with disease-modifying anti-rheumatic drugs or biological agents.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Kurimoto, MD, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ito Y, Hozumi K, Okada Y, Kurimoto S. Adalimumab with Methotrexate in Treatment-Naive Japanese Patients with Rheumatoid Arthritis at Risk of Progressive Structural Joint Damage: A Postmarketing Observational Study. Rheumatol Ther. 2017 Jun;4(1):151-166. doi: 10.1007/s40744-017-0059-1. Epub 2017 Mar 31. PMID 28364381
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who received adalimumab treatment
Period: Overall Study
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Started | 163
Completed | 157
Not Completed | 6
Not completed — Failed to meet inclusion criteria | 6

BASELINE CHARACTERISTICS:
Population: Participants who received adalimumab treatment
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient which does not necessarily have a causal relationship with their treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product. Adverse events were collected from the time of informed consent until the completion of the study, up to 26 weeks.
Time Frame: From baseline through week 26
Population: Participants who received adalimumab treatment
Measure: Number; unit: participants
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 157
participants | 40

2. Secondary Outcome: Mean Disease Activity Score 28 (DAS28-4(ESR)) at Baseline
Description: The DAS28-4(ESR) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR), and general health were included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: at week 0
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 121
units on a scale | 5.61 (1.39)

3. Secondary Outcome: Mean Disease Activity Score 28 (DAS28-4(ESR)) at Week 4
Description: The DAS28-4(ESR) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR), and general health were included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission .
Time Frame: at week 4
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 107
units on a scale | 3.57 (1.52)

4. Secondary Outcome: Mean Disease Activity Score 28 (DAS28-4(ESR)) at Week 12
Description: as for outcome 3
Time Frame: at week 12
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 90
units on a scale | 2.96 (1.35)

5. Secondary Outcome: Mean Disease Activity Score 28 (DAS28-4(ESR)) at Week 24
Description: as for outcome 2
Time Frame: at week 24
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 79
units on a scale | 2.41 (1.06)

6. Secondary Outcome: Percentage of Participants Achieving DAS28-4(ESR) Remission
Description: The DAS28-4(ESR) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR), and general health were included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. The percentage of participants with a DAS28 score <2.6 was documented.
Time Frame: From baseline to 24 weeks
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 131
percentage of participants
  Baseline, n=121 | 0.0
  Week 4, n=107 | 29.9
  Week 12, n=90 | 45.6
  Week 24, n=79 | 60.8

7. Secondary Outcome: Mean Clinical Disease Activity Index (CDAI) Score at Baseline
Description: The CDAI is a validated measure of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global health assessed by the participant on a visual analogue scale from 0 to 10 (cm), and global health assessed by an investigator on a visual analogue scale from 0 to 10 (cm) were included in the CDAI score. Scores on the CDAI range from 0 to 76. A CDAI score ≥22.1 indicates high disease activity, a CDAI score between 10.1 and 22.0 indicates moderate disease activity, a CDAI score between 2.9 and 10.0 indicates low disease activity, and a CDAI score ≤2.8 indicates clinical remission.
Time Frame: at week 0
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 138
units on a scale | 29.18 (14.38)

8. Secondary Outcome: Mean Clinical Disease Activity Index (CDAI) Score at Week 4
Description: as for outcome 7
Time Frame: at week 4
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 130
units on a scale | 10.95 (9.30)

9. Secondary Outcome: Mean Clinical Disease Activity Index (CDAI) Score at Week 12
Description: as for outcome 7
Time Frame: at week 12
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 108
units on a scale | 7.26 (7.73)

10. Secondary Outcome: Mean Clinical Disease Activity Index (CDAI) Score at Week 24
Description: as for outcome 7
Time Frame: at week 24
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 88
units on a scale | 3.96 (4.39)

11. Secondary Outcome: Percentage of Participants Achieving CDAI Remission
Description: The CDAI is a validated measure of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global health assessed by the participant on a visual analogue scale from 0 to 10 (cm) , and global health assessed by an investigator on a visual analogue scale from 0 to 10 (cm) were included in the CDAI score. Scores on the CDAI range from 0 to 76. A CDAI score ≥22.1 indicates high disease activity, a CDAI score between 10.1 and 22.0 indicates moderate disease activity, a CDAI score between 2.9 and 10.0 indicates low disease activity, and a CDAI score ≤2.8 indicates clinical remission. The percentage of participants with a CDAI score ≤2.8 was documented.
Time Frame: From baseline to 24 weeks
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 146
percentage of participants
  Baseline, n=138 | 0.7
  Week 4, n=130 | 20.0
  Week 12, n=108 | 35.2
  Week 24, n=88 | 60.2

12. Secondary Outcome: Mean Simplified Disease Activity Index (SDAI) Score at Baseline
Description: The SDAI is a validated measure of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global disease activity assessed by the participant on a visual analogue scale from 0 to 10 (cm) , global disease activity assessed by an investigator on a visual analogue scale from 0 to 10 (cm), and serum levels of C-reactive protein (mg/dL) were included in the SDAI score. Scores on the SDAI range from 0 to 86. An SDAI score ≥26.1 indicates high disease activity, an SDAI score between 11.1 and 26.0 indicates moderate disease activity, an SDAI score between 3.4 and 11.0 indicates low disease activity, and an SDAI score ≤3.3 indicates clinical remission.
Time Frame: at week 0
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 131
units on a scale | 32.30 (16.07)

13. Secondary Outcome: Mean Simplified Disease Activity Index (SDAI) Score at Week 4
Description: as for outcome 12
Time Frame: at week 4
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 123
units on a scale | 12.06 (10.20)

14. Secondary Outcome: Mean Simplified Disease Activity Index (SDAI) Score at Week 12
Description: as for outcome 12
Time Frame: at week 12
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 103
units on a scale | 8.08 (9.09)

15. Secondary Outcome: Mean Simplified Disease Activity Index (SDAI) Score at Week 24
Description: as for outcome 12
Time Frame: at week 24
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 85
units on a scale | 4.58 (4.93)

16. Secondary Outcome: Percentage of Participants Achieving SDAI Remission
Description: The SDAI is a validated measure of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global disease activity assessed by the participant on a visual analogue scale from 0 to 10 (cm) , global disease activity assessed by an investigator on a visual analogue scale from 0 to 10 (cm), and serum levels of C-reactive protein (mg/dL) were included in the SDAI score. Scores on the SDAI range from 0 to 86. An SDAI score ≥26.1 indicates high disease activity, an SDAI score between 11.1 and 26.0 indicates moderate disease activity, an SDAI score between 3.4 and 11.0 indicates low disease activity, and an SDAI score ≤3.3 indicates clinical remission. The percentage of participants with an SDAI score ≤3.3 was documented.
Time Frame: From baseline to 24 weeks
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Number analyzed (Participants) | 143
percentage of participants
  Baseline, n=131 | 0.0
  Week 4, n=123 | 22.0
  Week 12, n=103 | 39.8
  Week 24, n=85 | 58.8

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the time of informed consent until the last dose of adalimumab, up to 26 weeks.
Arm/Group | Participants With High Rheumatoid Arthritis Disease Activity
Serious Adverse Events (participants affected / at risk) | 4/157
Other Adverse Events (participants affected / at risk) | 36/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With High Rheumatoid Arthritis Disease Activity (N=157)
Pyelonephritis (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pericarditis (Cardiac disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With High Rheumatoid Arthritis Disease Activity (N=157)
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Dysphoria (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Liver disorder (Hepatobiliary disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site reaction (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Unevaluable event (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 1
Liver function test abnormal (Investigations) | 4
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 3
Blood beta-D-glucan increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Hepatic enzyme abnormal (Investigations) | 1
Mycobacterium tuberculosis complex test positive (Investigations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.